CLINICAL TRIAL: NCT00229801
Title: Evaluation of Renal Function in Children With Brain Tumors
Brief Title: Evaluation of Kidney Function in Children With Brain Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funds available, hard to enroll patients-Terminated in 2008
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Damian Grattan-Smith, MD, Children's Healthcare of Atlanta
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Renal Function/Brain Tumors
Record Dates: First submitted 2005-09-13; First posted 2005-09-30 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Brain Tumor
Keywords: Renal Function, MRI
MeSH Terms: conditions — Brain Neoplasms

ARMS (1):
- MRI (No Intervention)
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI

SUMMARY:
Clinical measurement of renal function is generally performed using either laboratory tests or nuclear medicine techniques, however, both of these techniques suffer from some limitations. Notably the lab tests only assess global, rather than individual kidney, function and the nuclear medicine tests are demanding to perform well. Children with brain tumors are often treated with chemotherapeutic in order to try and kill the cancer. Amongst the known side effect of some of the drugs used in the chemotherapy is the fact that they may damage the kidneys. For this reason the function of the kidneys is assessed using a laboratory test at 3 or 6 months intervals during the treatment. In addition, to the problem mentioned above the tests also require a separate visit to the hospital. Children with brain tumors who are undergoing chemotherapy also routinely have contrast-enhanced MRI of the brain performed at intervals of three months in order to evaluate the response of the tumor to the chemotherapy. Recently, MRI techniques have been developed which can evaluate single kidney renal function. The aim of this study is to establish if a single MRI exam can be used to assess both the effect of the chemotherapy on both the tumor and the renal function. The results of the MRI measurement of the single kidney renal function would be combined to provide a measure of global renal function and this would be compared with that obtained from the laboratory test. The MRI exam will require only require an extra 10 minutes of scanning time and will not affect the rest of the MRI exam in any way.

This study is being performed to validate a new technique for measuring kidney function. Patients are being asked to volunteer for this study because they require serial contrast enhanced MR scans to monitor their response to chemotherapy. Because some chemo-therapeutic agents can be toxic to the kidney the patient's kidney function will also be evaluated using conventional methods, and the results of these tests can be compared to those obtained using MRI. We plan to study 50 children in this study. The additional procedure for measuring renal function will add 10 minutes to the duration of the MRI exam and will have no effect on the routine brain study. If validated the proposed MRI technique would allow renal function to be evaluated at the time of a routine, contrast enhanced MRI exam and would avoid additional testing using radioactive tracers or urine collection over 24 hours.

If successful, MRI could be used to measure single kidney renal function in all any patient undergoing a routine MRI exam by simply extending the scanning time by a maximum of 10 minutes. This would save such patients additional visits to the hospital and would have the advantage of measuring single kidney, rather than global, renal function.

ELIGIBILITY:
Inclusion Criteria:

* All children currently enrolled, and who will be enrolled during the course of the study, in the chemotheraphy program at Children's Healthcare of Atlanta at Scottish Rite

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2004-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damien Grattan-Smith, MBBS, Principal Investigator — Children's Diagnostic Imaging of Atlanta/Children's Healthcare of Atlanta; Richard Jones, PhD, Principal Investigator — Emory University/Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia, United States